CLINICAL TRIAL: NCT03584113
Title: Video Assisted Thoracoscopic Decortication Versus Interventional Radiology Guided Chest Tube Insertion With Fibrinolytics for the Management of Empyema (DICE Trial)
Brief Title: VATS Decortication Versus IR Guided Chest Tube Insertion With Fibrinolytics for the Management of Empyema
Acronym: DICE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Wiley Chung (Other)
Responsible Party: Sponsor-Investigator, Dr. Wiley Chung, Principal Investigator, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6023903
Record Dates: First submitted 2018-06-17; First posted 2018-07-12 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Empyema, Pleural
MeSH Terms: conditions — Empyema, Pleural

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IR guided chest tube insertion with fibrinolytics (Active Comparator): Image guided chest tube insertion by interventional radiology along with MIST 2 trial fibrinolysis which includes intrapleural dornase (5mg) and Alteplase (10mg) every twelve hours for a total of six doses as primary intervention for empyema.
  Interventions: Other: Interventional radiology guided chest tube insertion with MIST2 trial fibrinolytics
- VATS Decortication (Active Comparator): Video assisted thorascopic surgery decortication (VATS) as primary intervention for empyema.
  Interventions: Other: Video assisted thorascopic decortication

INTERVENTIONS:
Other: Video assisted thorascopic decortication — Video assisted thorascopic decortication surgery as primary intervention for empyema
  Other Names: VATS Decortication
  Arms: VATS Decortication
Other: Interventional radiology guided chest tube insertion with MIST2 trial fibrinolytics — Image guided chest tube insertion by IVR with intrapleural fibrinolytics (six doses of dornase [5mg] and alteplase [10mg] Q12hours).
  Arms: IR guided chest tube insertion with fibrinolytics

SUMMARY:
The American Association of Thoracic Surgery defines empyema as pus in the pleural space. It is a common thoracic surgery presentation with an estimated 65,000 cases occurring annually in the United States. Despite the high prevalence of empyemas, there has been no consensus as to its optimal first line management. Methods of acceptable treatment currently include chest tube insertion (thoracostomy), thoracostomy with fibrinolytics, decortication via a thoracotomy (removal of fibrous peel on the lung) and video-assisted thoracoscopic surgery (VATS) decortication. The investigators aim to determine the rate of re-intervention within thirty days for adults presenting with empyema in the fibrinopurulent phase by comparing the initial treatments of Interventional Radiology (IR) guided chest tube insertion with intrapleural fibrinolytics (as per Multi-Institutional Sepsis 2 Trial; MIST 2 Trial) versus VATS decortication. Currently, either of these treatments is considered first-line depending on the surgeon and institutional preference.

DETAILED DESCRIPTION:
2.0 BACKGROUND INFORMATION AND RATIONALE

The European Association of Cardiothoracic Surgeons expert consensus statement for the surgical management of empyema groups empyema into three entities. They are Parapneumonic (stage I), Fibrinopurulent (Stage II) and Chronic Organizing (Stage III). Fibrinopurulent is further characterized by bacterial invasion across the damaged lung epithelium with pH<7.2, glucose <2.2mmol/L and LDH >1000IU/L. These criteria along with a positive culture, gram stain or observed pus, is defined as an empyema.

Despite the high incidence of empyemas, there continues to be controversy regarding first line management. Conventional thoracostomy has evolved to include the addition of intrapleural fibrinolytics for those in the fibrinopurulent phase. Many different agents and combinations of fibrinolytics have been described in the literature, as well as optimal techniques for chest tube insertion. With respect to fibrinolytics, the most recent MIST 2 randomized control trial (RCT) examined four separate treatment arms; double placebo, placebo combined with intrapleural DNAse (5mg), intrapleural t-PA (10mg) with placebo, and intrapleural t-PA (10mg) combined with DNase (5mg) for six doses over three days. This study demonstrated a statistically significant difference in the reduction of pleural empyema in the t-PA and DNase combined arm (P=0.005) when compared with all the other arms. This RCT has established intrapleural fibrinolytic therapy as the gold standard treatment for those with empyema. When considering thoracostomy itself, the literature overwhelmingly suggests that image-guided thoracostomy decreases the rate of complications (pneumothorax, infection, procedure failure, intercostal bleeding), compared with a blind chest tube insertion.

A Cochrane Systematic Review of eight trials (6 children and 2 adults) examining treatment methods for empyema provided moderate quality evidence suggesting there were similar complication rates between VATS decortication and chest tube drainage. The review also demonstrated VATS decortication potentially decreases hospitalization length of stay. A recent study examined 4,095 patients using the New York State database to investigate patients undergoing treatment for empyema with chest tube insertion, VATS decortication, or open thoracotomy. Patients had a higher mortality during their initial hospital stay when they received a chest tube compared with those who underwent a surgical approach (chest tube:15.4%, VATS:4.7%, open: 6.0%, p<0.001. Additionally, patients' readmission rate within thirty days was significantly higher for the chest tube group (6.1%) compared with the surgical group (VATS 1.9% and open: 2.1%, p<0.001) lending support that an initial surgical approach for empyema may be warranted.

Two separate adult RCTs have attempted to compare VATS decortication to thoracostomy with fibrinolytics. Wait et al. in 1997 used a small study population of twenty patients in each arm, randomizing participants to either bedside thoracostomy with streptokinase or VATS decortication. This study demonstrated that in adults with a fibrinopurulent effusion, VATS decortication is associated with an increased rate of empyema resolution and a shorter length of stay. A review article published by Chambers et al examined twenty-eight studies, comparing decortication via thoracotomy to VATS decortication for empyema. The majority of studies demonstrated that VATS has a decreased length of hospital stay, decreased postoperative morbidity and decreased post-operative pain. Furthermore, there was a higher resolution of empyema during the fibrinopurulent phase. Despite these two studies demonstrating superior outcomes with VATs decortication, they still do not compare modern day standards of treatment for empyema.

As the above literature suggests, there have been multiple proposed methods for first-line treatment of an empyema. However, there have not been any studies that compare modern standards of practice. Image-guided chest tube insertion has been shown to be superior to bedside chest tube insertion. Fibrinolytics administered as per MIST2 protocol has become the standard of practice at many institutions. Furthermore, VATS decortication has shown promising outcomes as first-line treatment and is associated with decreased morbidity compared with an open thoracotomy approach. Therefore, it is being proposed to compare image-guided chest tube insertion with MIST 2 trial fibrinolytics (six treatments of DNAse 5mg and t-PA 10mg over three days) to VATS decortication for the primary treatment of adults presenting with empyema in the fibrinopurulent phase. The investigators will determine the rate of re-intervention required within thirty days of treatment.

3.0 RESEARCH STUDY DESIGN/ METHODOLOGY This is a randomized control trial occurring at the Kingston Health Sciences Centre (KHSC). Empyema is a disease that is best managed with the expertise at an institution with thoracic surgeons. The standard practice is that once the diagnosis is made at another hospital in our LHIN, these patients are transferred to our Thoracic Surgery centre.

Patients will receive a baseline CT Chest to confirm the presence of an empyema. Participants will have a diagnostic pleural thoracentesis performed by their primary care team initially to determine whether the pleural fluid is an exudate suggestive of an empyema in its fibrinopurulent phase (see inclusion criteria). Once this is performed and the diagnosis of an empyema is obtained, patients in our LHIN not at KHSC will be transferred as usual to KHSC to be managed by the thoracic surgery team. For patients under the care of a different service at KHSC, they will be transferred to be under the care of the thoracic surgery team.

Once admitted under the thoracic surgery service, the study team will be notified and information will be provided to the patients. Informed consent will be obtained at this time by a member of the study team. Using an online randomization tool, participants will be randomized into either the image-guided thoracostomy combined with MIST 2 Trial fibrinolytics arm or the VATS decortication arm. Both procedures will be carried out within forty-eight hours of participant arrival. Both arms will also receive concurrent IV broad-spectrum antibiotics. The image-guided thoracostomy arm will go to the interventional radiology suite where a 12-24Fr chest tube will be inserted at the discretion of the interventional radiologist based on the specific clinical picture. Data will be collected during their stay. The primary outcome of the study will be to determine the rate of reintervention required, including additional chest tube insertion or surgery. Secondary outcomes will include mortality, duration of hospital stay, and adverse events. Data will be collected 30 days after their initial intervention to determine if any re-intervention was necessary.

A repeat CT Chest will be performed prior to discharge, clinical consideration of chest tube removal, or if there is no clinical improvement.

ELIGIBILITY:
Inclusion Criteria:

* CT Chest confirming the presence of a parapneumonic effusion
* Diagnostic thoracentesis values: pH<7.2, Glucose <2.2mmol/L or LDH >1000IU/L with the presence of pus
* Ability to undergo general anesthesia, no allergies to anesthetic agents or DNAse/streptokinase, no rapidly fatal underlying illness and the ability to tolerate single lung ventilation

Exclusion Criteria:

* Younger than age 18
* Pregnant
* Symptoms for six weeks or longer with a pleural peel on CT chest of ≥ 10mm thick as this would preclude patients to be better managed by thoracotomy rather than VATS
* Exhibiting signs of shock (hypotension, altered mental state etc)
* Participants cannot participate in any other clinical trials during the trial period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-08-24 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Rate of re-intervention | Thirty Days
  Requiring chest tube (+/-repeat), VATs decortication (+/-repeat), or thoracotomy

SECONDARY OUTCOMES:
Morbidity | Thirty Days
  post-intervention/ hospital complications
Mortality | Thirty Days
  post-intervention/ Hospital mortality
Resolution of Empyema | Up to 24 weeks
  Time to resolution of empyema
Cost of Hospital Stay | Measure from time to presentation to hospital to time of discharge
  Total costs calculated during hospital stay as a measure of global hospital costs

CONTACTS AND LOCATIONS:
Overall Officials: Wiley Chung, MD, FRCSC, Principal Investigator — Queens University; Erin Williams, MD, Study Director — Queens University
Locations (1):
- Queen's University/Kingston Health Sciences Centre, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
All data collected will be kept and analyzed amongst the co-investigators

REFERENCES:
- [Background] Ahmed S, Azam H, Basheer I. Is open decortication superior to fibrinolytic therapy as a first line treatment in the management of pleural empyema? Pak J Med Sci. 2016 Mar-Apr;32(2):329-32. doi: 10.12669/pjms.322.9676. PMID 27182233
- [Background] Chambers A, Routledge T, Dunning J, Scarci M. Is video-assisted thoracoscopic surgical decortication superior to open surgery in the management of adults with primary empyema? Interact Cardiovasc Thorac Surg. 2010 Aug;11(2):171-7. doi: 10.1510/icvts.2010.240408. Epub 2010 May 3. PMID 20439299
- [Background] Corcoran JP, Psallidas I, Wrightson JM, Hallifax RJ, Rahman NM. Pleural procedural complications: prevention and management. J Thorac Dis. 2015 Jun;7(6):1058-67. doi: 10.3978/j.issn.2072-1439.2015.04.42. PMID 26150919
- [Background] Havelock T, Teoh R, Laws D, Gleeson F; BTS Pleural Disease Guideline Group. Pleural procedures and thoracic ultrasound: British Thoracic Society Pleural Disease Guideline 2010. Thorax. 2010 Aug;65 Suppl 2:ii61-76. doi: 10.1136/thx.2010.137026. No abstract available. PMID 20696688
- [Background] Rahman NM, Maskell NA, West A, Teoh R, Arnold A, Mackinlay C, Peckham D, Davies CW, Ali N, Kinnear W, Bentley A, Kahan BC, Wrightson JM, Davies HE, Hooper CE, Lee YC, Hedley EL, Crosthwaite N, Choo L, Helm EJ, Gleeson FV, Nunn AJ, Davies RJ. Intrapleural use of tissue plasminogen activator and DNase in pleural infection. N Engl J Med. 2011 Aug 11;365(6):518-26. doi: 10.1056/NEJMoa1012740. PMID 21830966
- [Background] Redden MD, Chin TY, van Driel ML. Surgical versus non-surgical management for pleural empyema. Cochrane Database Syst Rev. 2017 Mar 17;3(3):CD010651. doi: 10.1002/14651858.CD010651.pub2. PMID 28304084
- [Background] Scarci M, Abah U, Solli P, Page A, Waller D, van Schil P, Melfi F, Schmid RA, Athanassiadi K, Sousa Uva M, Cardillo G. EACTS expert consensus statement for surgical management of pleural empyema. Eur J Cardiothorac Surg. 2015 Nov;48(5):642-53. doi: 10.1093/ejcts/ezv272. Epub 2015 Aug 7. PMID 26254467
- [Background] Semenkovich TR, Olsen MA, Puri V, Meyers BF, Kozower BD. Current State of Empyema Management. Ann Thorac Surg. 2018 Jun;105(6):1589-1596. doi: 10.1016/j.athoracsur.2018.02.027. Epub 2018 Mar 14. PMID 29550205
- [Background] Shen KR, Bribriesco A, Crabtree T, Denlinger C, Eby J, Eiken P, Jones DR, Keshavjee S, Maldonado F, Paul S, Kozower B. The American Association for Thoracic Surgery consensus guidelines for the management of empyema. J Thorac Cardiovasc Surg. 2017 Jun;153(6):e129-e146. doi: 10.1016/j.jtcvs.2017.01.030. Epub 2017 Feb 4. No abstract available. PMID 28274565
- [Background] Wait MA, Sharma S, Hohn J, Dal Nogare A. A randomized trial of empyema therapy. Chest. 1997 Jun;111(6):1548-51. doi: 10.1378/chest.111.6.1548. PMID 9187172